CLINICAL TRIAL: NCT04805502
Title: Effect of Exercise Modality During Pregnancy on Childhood Obesity Risk
Brief Title: Pregnancy Exercise Mode Effect on Childhood Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Linda May, Associate Professor; Interim Dept. Chair, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 19-001863
Record Dates: First submitted 2021-03-03; First posted 2021-03-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pregnancy; Overweight and Obesity
Keywords: exercise modes, exercise intervention
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: PRegnant women will be randomized to one of four groups: aerobic exercise, resistance exercise, combination (aerobic + resistance), or control (no exercise). All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, rating of perceived exertion (RPE), 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: those performing measurements on participants will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Aerobic Exercise (AE) (Experimental): All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, RPE, 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data.
  The AE group will exercise on aerobic machines (i.e. treadmill, elliptical, bicycle) for all of their sessions.
  Interventions: Behavioral: Exercise Modes
- Resistance Exercise (RE) (Experimental): All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, RPE, 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data.
  The RE group will perform 12-15 repetitions of 10-12 resistance exercises in a circuit, for 3 sets with rest period of 30-60 seconds between sets as needed.[100] Seated isokinetic exercise using Cybex machines will target all major muscle groups. Light dumbbells and resistance bands will be used if the participant is unable to lift the minimal load on Cybex machines. Core exercises will be performed at the end of the session (i.e. seated side bends).
  Interventions: Behavioral: Exercise Modes
- Combination Exercise (AERE) (Experimental): All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, RPE, 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data.
  The AERE group will switch between AE exercise and RE; for this group, RE exercises will consist of 1 set of 12-15 repetitions of 4 resistance exercises, then 5 minutes of AE, then repeated repeat with different exercises.[106-108] The investigators will also calculate the metabolic minutes per week (METmin/wk) of all participants in order to account for potential differences in energy expenditure based on activity, though the dose of 150 min/wk at moderate intensity is held constant between exercise groups.
  Interventions: Behavioral: Exercise Modes
- Control (no exercise) (No Intervention): The Control group will participate in weekly sessions that focus on stretching, breathing, and healthy lifestyle.

INTERVENTIONS:
Behavioral: Exercise Modes — Moderate intensity aerobic exercise, moderate intensity resistance exercise, moderate intensity combination exercise
  Arms: Aerobic Exercise (AE); Combination Exercise (AERE); Resistance Exercise (RE)

SUMMARY:
The overall objective of this proposal is to conduct a longitudinal prospective study of overweight/obese (OW/OB) pregnant women and their offspring to determine which prenatal exercise mode will have the greatest impact on maternal and infant cardiometabolic health. This information may lead to clinical practice recommendations that improve childhood health. This randomized controlled trial will recruit 284 OW/OB pregnant women randomized to an exercise intervention (aerobic (AE), resistance (RE), or aerobic+resistance exercise (AERE)) or to no exercise; their infants will be measured at 1, 6, and 12 months of age. This design will test our central hypothesis that AERE and RE training during pregnancy will improve maternal and offspring cardiometabolic outcomes to a greater extent than AE alone. This hypothesis will be tested with two specific aims:

Aim 1. Determine the influence of different exercise modes during OW/OB pregnancy on infant cardiometabolic health and growth trajectories. Hypothesis: AE, RE, and AERE by OW/OB pregnant women will improve offspring neuromotor and cardiometabolic measures at 1, 6, and 12 months postpartum (e.g. decreased %body fat, BMI z-score, heart rate [HR], non-HDL, and C-Reactive Protein (CRP); increased insulin sensitivity) compared to infants of OW/OB pregnant women that do not exercise; AERE and RE will have the greatest impact on improving infant measures.

Aim 2. Determine the most effective exercise mode in OW/OB pregnancy on improving maternal cardiometabolic health outcomes. Hypothesis: AE, RE, and AERE by OW/OB pregnant women will improve both maternal cardiometabolic health measures (e.g. decreased BMI z-score, non-HDL, % body fat, HR, weight gain) across pregnancy (16-36 weeks' gestation) and overall pregnancy outcomes (e.g. lower incidence of gestational diabetes, pre-eclampsia, hypertension during gestation) compared to OW/OB pregnant women that do not exercise; AERE and RE will have the greatest impact on improving maternal health measures, with the AERE group having the highest compliance.

The proposed study will be the first to provide an understanding of the influence of maternal exercise modes on the cardiometabolic health and growth trajectories of offspring who are at increased risk due to maternal OW/OB. This work will have a significant impact on reducing the cycle of OB, potentially providing the earliest and most efficacious intervention to decrease or prevent OB in the next generation.

DETAILED DESCRIPTION:
Many public health initiatives in the United States, including Healthy People 2020, have goals that include reducing obesity (OB), metabolic dysfunction, and risk of cardiovascular disease (CVD). Studies such as the Bogalusa project have now demonstrated that overweightness (OW), beginning as early as age five, is predictive of adult CVD. In fact, the onset of OW/OB and CVD may begin in the intrauterine period, and infant birth weight and weight gain are strongly related to OB in childhood and beyond. OW/OB mothers and their offspring exhibit increased morbidity and mortality; the American College of Obstetricians and Gynecologists (ACOG) has developed guidelines geared toward reducing maternal OW/OB through exercise. However, few studies have focused on how such exercise interventions during pregnancy impact short and long-term child health outcomes. Furthermore, little is known regarding the influence of different modes of antenatal exercise upon maternal and offspring health outcomes.

The long-term goal of this study is to attenuate child- and adulthood OB and CVD risk by identifying the most effective and easily implemented maternal exercise interventions. The investigators have shown that maternal aerobic exercise (AE) in women of all BMIs favorably impacts maternal cholesterol and LDL levels, which are predictive of infant weight. Furthermore, maternal AE is associated with decreased fetal abdominal circumference (AC), lower body fat percentage at one month, and improved infant neuromotor skills. Our preliminary data for pregnant women of all BMIs suggests that resistance exercise (RE) confers similar benefits to infants at one month as compared to AE, plus improvements such as decreased BMI z-scores, increased metabolomic signatures for glucose use, and decreased metabolites of inflammatory pathways. The most striking finding from this preliminary work is that adding RE to AE improved outcomes for both mothers and infants. Thus, the COMBINATION of aerobic and resistance exercise (AERE) not only had better maternal and one month infant outcomes (versus AE alone), but AERE groups had the best compliance. The positive changes were most pronounced in the infants of OW/OB women. A more comprehensive, longitudinal study geared toward OW/OB mothers is needed to confirm our preliminary work and to assess the persistence of exercise impacts through the infants' first year of life.

The overall objective of this proposal is to conduct a longitudinal prospective study of OW/OB pregnant women and their offspring to determine which antenatal maternal exercise mode(s) will have the greatest impact on maternal and infant cardiometabolic health. This information may lead to modified clinical practice recommendations that improve health in childhood and possibly beyond. This randomized controlled trial will recruit 284 OW/OB pregnant women randomized to an exercise intervention (AE, RE, AERE) or to no exercise (usual care); their infants will be measured at 1, 6, and 12 months of age. This rigorous design will test our central hypothesis that AERE and RE exercise training during pregnancy will, in OW/OB women, improve maternal and offspring cardiometabolic outcomes to a greater extent than AE alone. The investigators will test this hypothesis with two specific aims:

Aim 1. Determine the influence of different exercise modes during OW/OB pregnancy on infant cardiometabolic health and growth trajectories. Hypothesis: AE, RE, and AERE by OW/OB pregnant women will improve offspring neuromotor and cardiometabolic measures at 1, 6, and 12 months postpartum (e.g. decreased BMI z-score, body fat %, non-HDL, heart rate, and C-Reactive Protein (CRP); increased insulin sensitivity) compared to infants of OW/OB pregnant women that do not exercise; AERE and RE will have the greatest impact on improving infant measures.

Aim 2. Determine the most effective exercise mode in OW/OB pregnancy on improving maternal cardiometabolic health outcomes. Hypothesis: AE, RE, and AERE by OW/OB pregnant women will improve both maternal cardiometabolic health measures (e.g. decreased BMI z-score, body fat %, HR, non-HDL, weight gain) across pregnancy (~13 to ~40 weeks gestation) and overall pregnancy outcomes (e.g. lower incidence of gestational diabetes, pre-eclampsia, hypertension during gestation) compared to OW/OB pregnant women that do not exercise; AERE and RE will have the greatest impact on improving maternal health measures, with the AERE group having the highest compliance with improved health outcomes.

The proposed innovative study will be the first to provide a critical understanding of the influence of antenatal exercise modes upon the cardiometabolic health and growth trajectories of offspring who are at increased risk due to maternal OW/OB. This work will have a significant impact on reducing the cycle of OB and CVD, potentially providing the earliest and most efficacious intervention to attenuate or prevent OB and CVD in the next generation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 40 years old
* BMI between ≥ 25
* Pregnancy: Singleton; ≤ 16 weeks gestation
* Clearance by Obstetric provider for exercise

Exclusion Criteria:

* Age: ≤ 17.9 or ≥ 41 years of age
* BMI <25
* Multi fetal pregnancy
* Obstetric Provider does not provide clearance for exercise
* Unable or Unwilling to provide consent
* Inability to communicate with members of study team, despite use of interpreter
* Medical Conditions (e,g. HIV/Aids, Cancer, Type 1 or 2 Diabetes, Untreated Hypertension, Thyroid Disorders)
* Use of tobacco products, alcohol, recreational drugs, or medications (oral hypertensive, insulin)
* Unable to provide phone or email contact

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
1 month Infant non-HDL | 1 month
  non-HDL measured from venipuncture
6 month Infant non-HDL | 6 months
  non-HDL measured from venipuncture
12 month Infant non-HDL | 12 months
  non-HDL measured from venipuncture
1 month Infant BMI z-score | 1 month
  BMI normalized
6 month Infant BMI z-score | 6 months
  BMI normalized
12 month Infant BMI z-score | 12 months
  BMI normalized
Enrollment (8-13wks) Maternal fasting non-HDL | enrollment (~8-13 wks gestation)
  non-HDL measured from venipuncture
36wk Maternal fasting non-HDL | 36 weeks gestation
  non-HDL measured from venipuncture
1 month postpartum Maternal fasting non-HDL | 1 month postpartum
  non-HDL measured from venipuncture
6 months postpartum Maternal fasting non-HDL | 6 months postpartum
  non-HDL measured from venipuncture
Adverse Pregnancy Outcomes | At Delivery
  Presence or absence of Adverse Pregnancy outcomes (preterm birth, gestational diabetes [GDM], preeclampsia, hypertension)

SECONDARY OUTCOMES:
1 month Infant Resting Heart Rate | 1 month
  resting HR
6 month Infant Resting Heart Rate | 6 months
  resting HR
12 month Infant Resting Heart Rate | 12 months
  resting HR
1 month Infant Resting Blood Pressure | 1 month
  resting BP
6 month Infant Resting Blood Pressure | 6 months
  resting BP
12 month Infant Resting Blood Pressure | 12 months
  resting BP
1 month Infant Body Fat % | 1 month
  estimated body fat % from skinfolds
6 month Infant Body Fat % | 6 months
  estimated body fat % from skinfolds
12 month Infant Body Fat % | 12 months
  estimated body fat % from skinfolds
1 month Infant % Muscle Mass | 1 months
  estimated muscle mass % from skinfolds
6 month Infant % Muscle Mass | 6 months
  estimated muscle mass % from skinfolds
12 month Infant % Muscle Mass | 12 months
  estimated muscle mass % from skinfolds
1 month Infant Resting Energy Expenditure (REE) | 1 months
  estimated REE
6 month Infant Resting Energy Expenditure (REE) | 6 months
  estimated resting energy expenditure
12 month Infant Resting Energy Expenditure (REE) | 12 months
  estimated resting energy expenditure
1 month Infant Neuromotor Assessment | 1 months
  Peabody Developmental Motor Scale (1st - 99th percentile) - the higher the percentile the better
6 month Infant Neuromotor Assessment | 6 months
  Peabody Developmental Motor Scale (1st - 99th percentile) - the higher the percentile the better
12 month Infant Neuromotor Assessment | 12 months
  Peabody Developmental Motor Scale (1st - 99th percentile) - the higher the percentile the better
1 month Infant Veggie Meter | 1 month
  Raman Spectroscopy-Skin Carotenoid assessments
6 month Infant Veggie Meter | 6 months
  Raman spectroscopy-Skin Carotenoid assessments
12 month Infant Veggie Meter | 12 months
  Raman spectroscopy-Skin Carotenoid assessments
1 month Infant Blood Biomarkers (CRP) | 1 month
  Multiplex analyses of inflammatory markers (CRP)
6 month Infant Blood Biomarkers (CRP) | 6 months
  Multiplex analyses of inflammatory markers (CRP)
12 month Infant Blood Biomarkers (CRP) | 12 months
  Multiplex analyses of inflammatory markers (CRP)
1 month Infant Blood Biomarkers (IL6) | 1 month
  Multiplex analyses of inflammatory markers (IL6)
6 month Infant Blood Biomarkers (IL6) | 6 months
  Multiplex analyses of inflammatory markers (IL6)
12 month Infant Blood Biomarkers (IL6) | 12 months
  Multiplex analyses of inflammatory markers (IL6)
1 month Infant Blood Biomarkers (adiponectin) | 1 month
  Multiplex analyses of inflammatory markers (adiponectin)
6 month Infant Blood Biomarkers (adiponectin) | 6 month
  Multiplex analyses of inflammatory markers (adiponectin)
12 month Infant Blood Biomarkers (adiponectin) | 12 months
  Multiplex analyses of inflammatory markers (adiponectin)
1 month Infant Metabolomics | 1 month
  Metabolomic pathway analysis of significantly different blood metabolites based on p-value less than or equal to 0.05
6 month Infant Metabolomics | 6 months
  Metabolomic pathway analysis of significantly different blood metabolites based on p-value less than or equal to 0.05
12 months Infant Metabolomics | 12 months
  Metabolomic pathway analysis of significantly different blood metabolites based on p-value less than or equal to 0.05
16wk Maternal Resting Heart Rate | 16 gestation
  resting HR
36wk Maternal Resting Heart Rate | 36 weeks gestation
  resting HR
1 month postpartum Maternal Resting Heart Rate | 1 month postpartum
  resting HR
6 month postpartum Maternal Resting Heart Rate | 6 months postpartum
  resting HR
16wk Maternal Resting Blood Pressure | 16 weeks gestation
  resting BP
36wk Maternal Resting Blood Pressure | 36 weeks gestation
  resting BP
1 month postpartum Maternal Resting Blood Pressure | 1 month postpartum
  resting BP
6 month postpartum Maternal Resting Blood Pressure | 6 months postpartum
  resting BP
Maternal Gestational Weight Gain (GWG) | at delivery
  Gestational Weight Gain
16wk Maternal Body Fat% | 16 weeks gestation
  Estimated body fat %
36wk Maternal Body Fat% | 36 weeks gestation
  Estimated body fat %
1 month Postpartum Maternal Body Fat% | 1 month postpartum
  Estimated body fat %
6 month Postpartum Maternal Body Fat% | 6 months postpartum
  Estimated body fat %
16wk Maternal Biomarkers (CRP) | 16 weeks gestation
  Multiplex analyses of inflammatory markers (CRP)
36wk Maternal Biomarkers (CRP) | 36 weeks gestation
  Multiplex analyses of inflammatory markers (CRP)
1 month postpartum Maternal Biomarkers (CRP) | 1 month postpartum
  Multiplex analyses of inflammatory markers (CRP)
6 month Postpartum Maternal Biomarkers (CRP) | 6 months postpartum
  Multiplex analyses of inflammatory markers (CRP)
16wk Maternal Biomarkers (IL6) | 16 weeks gestation
  Multiplex analyses of inflammatory markers (IL6)
36wk Maternal Biomarkers (IL6) | 36 weeks gestation
  Multiplex analyses of inflammatory markers (IL6)
1 month Postpartum Maternal Biomarkers (IL6) | 1 month postpartum
  Multiplex analyses of inflammatory markers (IL6)
6 month Postpartum Maternal Biomarkers (IL6) | 6 months postpartum
  Multiplex analyses of inflammatory markers (IL6)
16wk Maternal Biomarkers (adiponectin) | 16 weeks gestation
  Multiplex analyses of inflammatory markers (adiponectin)
36wk Maternal Biomarkers (adiponectin) | 36 weeks gestation
  Multiplex analyses of inflammatory markers (adiponectin)
1 month Postpartum Maternal Biomarkers (adiponectin) | 1 month postpartum
  Multiplex analyses of inflammatory markers (adiponectin)
6 month Postpartum Maternal Biomarkers (adiponectin) | 6 months postpartum
  Multiplex analyses of inflammatory markers (adiponectin)
16wk Maternal Biomarkers (cortisol) | 16 weeks gestation
  Multiplex analyses of inflammatory markers (cortisol)
36wk Maternal Biomarkers (cortisol) | 36 weeks gestation
  Multiplex analyses of inflammatory markers (cortisol)
1 month Postpartum Maternal Biomarkers (cortisol) | 1 month postpartum
  Multiplex analyses of inflammatory markers (cortisol)
6 month Postpartum Maternal Biomarkers (cortisol) | 6 months postpartum
  Multiplex analyses of inflammatory markers (cortisol)

CONTACTS AND LOCATIONS:
Overall Officials: Linda E May, PhD, Principal Investigator — PI
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
de-identified data can be shared upon request to researchers

REFERENCES:
- [Derived] Jevtovic F, Wisseman BL, Jahan F, Claiborne A, Collier DN, DeVente JE, Mouro S, Zeczycki T, Szumilewicz A, Adamo KB, Goodyear LJ, May LE. Maternal exercise alters placental proteome in an exercise mode-specific manner. Am J Physiol Endocrinol Metab. 2025 Dec 1;329(6):E912-E922. doi: 10.1152/ajpendo.00052.2025. Epub 2025 Nov 4. PMID 41187954
- [Derived] Jevtovic F, Claiborne A, DeVente JE, Mouro S, Houmard JA, Broskey NT, May LE. Maternal resistance exercise increases infant energy expenditure. Am J Physiol Endocrinol Metab. 2025 Mar 1;328(3):E354-E361. doi: 10.1152/ajpendo.00414.2024. Epub 2024 Dec 23. PMID 39716848
- [Derived] Jevtovic F, Collier DN, DeVente J, Mouro S, Claiborne A, Wisseman B, Steen D, Kern K, Broskey N, May LE. Maternal exercise increases infant resting energy expenditure: preliminary results. Int J Obes (Lond). 2024 Sep;48(9):1347-1350. doi: 10.1038/s41366-024-01560-0. Epub 2024 Jun 10. PMID 38858465